CLINICAL TRIAL: NCT03806920
Title: Isomaltulose VS Sucrose - Different Postprandial Effect on Incretin Profile and Determinants of the Second Meal Effect
Brief Title: Isomaltulose VS Sucrose - Postprandial Effect on Incretin Profile and Second Meal Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Beneo GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director (Dpt. Clinical Nutrition), German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PALA
Record Dates: First submitted 2017-11-08; First posted 2019-01-16 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome
Keywords: Isomaltulose; Palatinose; second meal effect; incretin; GIP; GLP-1; postprandial inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Comparison of sucrose vs. palatinose (isomaltulose) on second meal effect (high-GI meal vs. high-protein meal) in subjects with T2DM or metabolic Syndrome without T2DM
Who Masked: Participant
Masking Description: participants were unaware of selected sugar intake prior to second meal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention A (Active Comparator): Nutritional intervention in healthy subjects and T2DM subjects:
  Accompanying a carbohydrate based breakfast, participants ingest either 50 g sucrose followed by a standardized lunch on 1 single day. In addition, blood samples are taken over 8 hours.
  Interventions: Dietary Supplement: Intervention A
- Intervention B (Active Comparator): Nutritional intervention in healthy subjects and T2DM subjects:
  Accompanying a carbohydrate based breakfast, participants ingest either 50 g palatinose followed by a standardized lunch on 1 single day. In addition, blood samples are taken over 8 hours.
  Interventions: Dietary Supplement: Intervention B
- Intervention C (Active Comparator): Nutritional intervention in healthy subjects:
  Accompanying a protein-based breakfast, participants ingest either 50 g sucrose followed by a standardized lunch on 1 single day. In addition, blood samples are taken over 8 hours.
  Interventions: Dietary Supplement: Intervention C
- Intervention D (Active Comparator): Nutritional intervention in healthy subjects:
  Accompanying a protein-based breakfast, participants ingest either 50 g isomaltulose followed by a standardized lunch on 1 single day. In addition, blood samples are taken over 8 hours.
  Interventions: Dietary Supplement: Intervention D

INTERVENTIONS:
Dietary Supplement: Intervention A
  Arms: Intervention A
Dietary Supplement: Intervention B
  Arms: Intervention B
Dietary Supplement: Intervention C
  Arms: Intervention C
Dietary Supplement: Intervention D
  Arms: Intervention D

SUMMARY:
This study evaluates the different postprandial effect of isomaltulose and sucrose on the incretin profile and as an determinant for the second meal effect.

In this nutritional intervention study, healthy participants and T2DM patients ingest 2 standardized meals for breakfast and lunch in combination with either sucrose or palatinose on 2 separate days. In addition, blood samples are taken to analyze markers of the carbohydrate metabolism, incretins and specific inflammation markers.

DETAILED DESCRIPTION:
Isomaltulose is a natural occurring disaccharide with a similar structure to sucrose. It is composed of glucose and fructose, but is linked by an α-1,6-glycosidic bond instead of α-1,2. Due to its binding, isomaltulose is slowly hydrolysed, which results in a rather weak postprandial glycemic-insulinemic response, accompanied by a minimal GIP secretion and a stimulated secretion of GLP-1. In addition, several studies have shown that the intake of foods with a low glycemic index, such as isomaltulose, tend to improve the metabolic reaction to a subsequent meal. As the exact mechanism of this "second meal effect" is still unknown, the investigators hypothesize that the modified release and action of GIP and GLP-1 are key players in regard to the described effects.Therefore, isomaltulose could be a suitable tool for reducing the risk of developing diabetes, obesity and CVD as well as improve blood glucose control in people with diabetes.

In summary, this study evaluates the different postprandial effect of isomaltulose and sucrose on the incretin profile and as a determinant for the second meal effect.

In this nutritional intervention study, healthy participants and T2DM patients ingest 2 standardized meals for breakfast and lunch in combination with either sucrose or palatinose on 2 separated days. In addition, blood samples are taken to analyze markers of the carbohydrate metabolism, incretins and specific inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* for T2DM patients: insulin-independent
* for healthy subjects: at least 1 component of the metabolic syndrom:

  * Body mass index (BMI) ≥ 30 kg/m²
  * Waist-hip ratio (WHR) ≥ 85 for women and ≥ 90 for men
  * hypertension
  * dyslipidemia
  * glucose / insulin intolerance

Exclusion Criteria:

* medications: intake of medications which influence glucose metabolism
* alcohol / drug abuse
* physical diseases: endocrinological, malign, serious cardiovascular diseases
* acute / chronic communicable disease
* psychic diseases

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-05 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
disposition index | 4 visits, separated by 1 week each
  Alteration of the Insulin secretion due to the intake of isomaltulose or sucrose in combination with different times and meal compositions. This should lead to an improved beta-cell response (Insulin secretion)
insulinogenic index | 4 visits, separated by 1 week each
  Alteration of the incretin profile due to the intake of isomaltulose or sucrose in combination with different times and meal compositions. This should lead to an improved second meal effect (Insulin sensitivity).
hepatic insulin extraction | 4 visits, separated by 1 week each
  Alteration of the incretin profile due to the intake of isomaltulose or sucrose in combination with different times and meal compositions. This should lead to an improved hepatic insulin extraction (secondary effect of improved Insulin sensitivity).

SECONDARY OUTCOMES:
incretin response | 4 visits, separated by 1 week each
  Parameters: GIP, GLP-1, gastric emptying, Glucagon
inflammatory reaction | 4 visits, separated by 1 week each
  Parameters: IL8, IL-18
Lipid status | 4 visits, separated by 1 week each
  Parameters: NEFA
additional endocrine parameters | 4 visits, separated by 1 week each
  Parameters: FGF21

CONTACTS AND LOCATIONS:
Locations (1):
- German Institute of Human Nutrition, Potsdam, Brandenburg, Germany

REFERENCES:
- [Derived] Zhang J, Schafer SM, Kabisch S, Csanalosi M, Schuppelius B, Kemper M, Markova M, Meyer NMT, Pivovarova-Ramich O, Keyhani-Nejad F, Rohn S, Pfeiffer AFH. Implication of sugar, protein and incretins in excessive glucagon secretion in type 2 diabetes after mixed meals. Clin Nutr. 2023 Apr;42(4):467-476. doi: 10.1016/j.clnu.2023.02.011. Epub 2023 Feb 21. PMID 36857956